CLINICAL TRIAL: NCT07081620
Title: How Long Does it Take for Percutaneous Intercostal Cryoneuromodulation to Produce Cryoanalgesia? A Prospective Observational Study.
Brief Title: Percutaneous Intercostal Cryoneuromodulation Onset Timing.
Status: Recruiting | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Stefano Mariconti, Principal Investigator, Papa Giovanni XXIII Hospital
Other Study IDs: PICOT1
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cryotherapy Effect; Pectus Excavatum
Keywords: Cryoneurolysis; Cryoneuromodulation
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pectus patients: Patients who are eligible for Nuss procedure (for pectus excavatum correction) are undergoing "earlier preoperative percutaneous intercostal cryoneurolysis" in our institution. They are studied through a physical examination also.
  Interventions: Other: Physical examination of chest skin

INTERVENTIONS:
Other: Physical examination of chest skin — soft touch and thermal (cold and warm) examination

SUMMARY:
Percutaneous Intercostal Cryoneurolysis is a promising technique that addresses acute postoperative pain after Nuss procedure for pectus excavatum. However its onset timing has not yet been determined. A physical examination would assess the variation of chest skin sensitivity to soft touch, cold (water at 4°C), and heat (water at 40°C) through days following the cryoneurolysis procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing preoperative percutaneous intercostal cryoneurolysis for pectus excavatum surgery

Exclusion Criteria:

* failure to obtain consent

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Mainly adolescents, mainly males
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
thermal sensitivity | one week (median)
  Chest skin thermal sensitivity will be assessed through a "thermofeel" metal instrument set at two different temperatures: 15°C for cold sensation and 40°C for warm sensation. At least 4 different chest zones will be tested to discriminate potential differences. As a validated instument for chest skin thermal assessment does not exist, we will report only qualitative results, as "normal" "impaired" or "absent" sensitivity.

SECONDARY OUTCOMES:
chest skin sensitivity to touch | one week (median)
  Chest skin mechanical sensitivity will be assessed through both validated von Frey filament testing, and cotton swab for soft touch. At least 4 different chest zones will be tested to discriminate potential differences. We will report qualitative results, as "normal" "impaired" or "absent" sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Papa Giovanni XXIII Hospital, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Population basic data

REFERENCES:
- [Background] Mariconti S, Bronco A, Pellicioli I, Chiudinelli L, Cattaneo M, Cheli M, Bonanomi E. Earlier preoperative percutaneous intercostal cryoanalgesia improves recovery after pectus excavatum surgery. Reg Anesth Pain Med. 2024 Nov 7:rapm-2024-105960. doi: 10.1136/rapm-2024-105960. Online ahead of print. PMID 39510802